CLINICAL TRIAL: NCT00411567
Title: An Open Label Study to Assess the Utility of Measuring Markers of Inflammation, to Detect Transition From Optimal to Sub-Optimal Inhaled Corticosteroid Therapy in Moderate-Severe Bronchial Asthma
Brief Title: A Study to Assess the Efficacy of Inhaled Corticosteroid (ICS) Therapy in Moderate-Severe Bronchial Asthma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQAE397A2202
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Bronchial Asthma
Keywords: markers, inflammation, optimal, sub-optimal, corticosteroid, bronchial asthma
MeSH Terms: conditions — Asthma; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: inhaled corticosteroid therapy

SUMMARY:
The purpose of this study is to investigate/assess the treatment of moderate to severe asthmatics with inhaled corticosteroid.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female moderate to severe asthmatic patients, from 18-75 years of age.
* Moderate to severe asthma, according to the GINA guidelines, for at least one year with no exacerbations requiring hospitalization and/or oral steroids within the previous three months.
* No concomitant lung disease or significant medical conditions
* Fluticasone propionate 500mcg daily or greater, or equivalent (Mometsaone 800 mcg, triamcinolone 2000 mcg, Flunisolide 2000 mcg, Budesonide DPI 800 mcg, Beclomathasone HFA 500 mcg, Beclomethasone CFC 1000 mcg, Forced expiratory volume in 1 second (FEV1) at screening will be ≥ 70% of the normal predicted.
* Evidence of asthma, demonstrated by one of the following: Historical evidence confirmed by their treating physician or Demonstration of ≥ 12% reversibility of FEV1 using a standard dose of salbutamol (up to 400 µg) within 30 minutes.
* Female subjects of child bearing potential must be using two forms of contraception or postmenopausal women must have no regular menstrual bleeding for at least 2 years prior to inclusion.
* Body Mass Index between 18 and 30. Body weight should be less than 100 kg.

Exclusion Criteria:

* Smokers
* Concomitant medications: Except for short- and long-acting β-agonists and medication which may be required to treat adverse events, all other medications, other than study drug should be avoided from screening until all of the study completion evaluations have been conducted. Paracetamol is acceptable.
* Medical conditions: history of clinically significant drug allergy; any significant medical condition. For example, a history of any pulmonary disorder other than asthma.
* Any surgical or medical condition which might significantly alter the distribution, metabolism or excretion of the drug.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing or longer if required by local regulation.
* Significant illness within the two weeks prior to dosing.
* A past personal or close family medical history of clinically significant cardiac abnormalities
* History of history of fainting, orthostatic hypotension, sinus arrhythmia, etc.
* A known hypersensitivity to Fluticasone propionate or drugs similar to Fluticasone propionate.
* History of immunocompromise, including a positive HIV test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of drug or alcohol abuse within the 12 months prior to dosing

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 2006-07

PRIMARY OUTCOMES:
Change in inflammatory parameters in response to a decrease in ICS compared to no change in therapy after 2 and 4 weeks

SECONDARY OUTCOMES:
Parameter/combination of parameters most sensitive to the ICS reduction
Collection of relative data to assess sample size calculations for subsequent studies

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Nuremberg, Germany